CLINICAL TRIAL: NCT05524688
Title: Yeast-derived Beta-glucan Supplementation for Fatigue Symptoms in Autologous Haemopoietic Stem Cell Transplant Survivors
Brief Title: Beta-glucan and Fatigue in HSCT Survivors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Departure of PI clinician from institution.
Sponsor: University of Florida (Other)
Collaborators: Lallemand Bio-Ingredients (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB202102622
Record Dates: First submitted 2022-08-30; First posted 2022-09-01 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Autologous Haemopoietic Stem Cell Transplant
Keywords: HSCT; fatigue; beta-glucan; quality of life; inflammation
MeSH Terms: conditions — Fatigue; Inflammation | interventions — beta-Glucans

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Beta-glucan (Experimental): 500 mg/d of beta-glucan
  Interventions: Dietary Supplement: Beta-glucan
- Placebo (Placebo Comparator): 500 mg/d of cellulose
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Beta-glucan — 2, 250 mg capsules of beta-glucan per day
  Arms: Beta-glucan
Dietary Supplement: Placebo — 2, 250 mg capsules of cellulose
  Arms: Placebo

SUMMARY:
This is a single-center, randomized, double-blind, placebo-controlled study exploring the effects of a yeast-derived β-glucan on clinically significant fatigue among survivors of autologous HCT due to multiple myeloma. The primary aim is to evaluate the effect of β-glucan supplementation on changes in fatigue symptoms, as assessed by the Brief Fatigue Inventory (BFI) global fatigue score, by testing the differences in changes in scores from baseline to the mid-point (mean of weeks 1-4) and to the end of the intervention (mean of weeks 5-8).

DETAILED DESCRIPTION:
Fatigue is one of the most prevalent and distressing complications among hematopoietic cell transplantation HCT survivors, affecting up to 80% of patients. Fatigue has a significant negative impact on the physical, functional, social, and emotional domains of quality of life. Therefore, special attention should be directed toward therapeutic interventions in reducing persistent fatigue, which in turn improves quality of life of this patient population. Research is needed to determine if yeast-derived β-glucan regulates inflammatory disruption and fatigue in patient populations. This study will investigate the efficacy of β-glucan supplementation on fatigue symptoms in autologous HCT survivors due to multiple myeloma. The primary aim is to evaluate the effect of β-glucan supplementation on changes in fatigue symptoms, as assessed by the BFI global fatigue score, by testing the differences in changes in scores from baseline to the mid-point (mean of weeks 1-4) and to the end of the intervention (mean of weeks 5-8). Secondary objectives will be to evaluate tolerability, adverse events, inflammatory cytokines, quality of life, sleep disturbance, pain, anxiety, and depression.

ELIGIBILITY:
Inclusion Criteria:

* Be ≥ 18 years of age.
* Be an autologous HSCT survivor with clinically significant fatigue (determined post-consent). Clinically significant fatigue is defined as BFI global score greater than 3.0.
* Have a medical history of the first autologous HSCT due to multiple myeloma approximately 30 days before starting the study intervention.
* Be willing and able to provide written informed consent.
* Be willing and able to comply with all the study-related procedures, including attending study visits for the blood draws, intake of the study supplement, and completing study questionnaires.

Exclusion Criteria:

* Have an active infection.
* Have disease relapse.
* Have absolute neutrophil count less than 500.
* Have anemia and thrombocytopenia requiring transfusions.
* Have an untreated medical condition that could clinically explain fatigue in this population (i.e., untreated hypothyroidism).
* Have begun to take antidepressants less than 30 days from enrollment.
* Demonstrate an inability to comply with the study and/or follow-up procedures.
* Use probiotic supplements. The subjects can participate if they are willing to stop taking probiotics. A one-month withdrawal from probiotics is required

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2023-02-10 (Actual); Primary Completion 2023-08-28 (Actual); Study Completion 2023-08-28 (Actual)

PRIMARY OUTCOMES:
Change in fatigue as assessed by Brief Fatigue Inventory (BFI) tool | 8 weeks
  change in global fatigue score

SECONDARY OUTCOMES:
Frequency of adverse events per group | 8 weeks
  number of adverse events
Change in serum levels of TNF-α, IL-1β, and IFN-γ | 8 weeks
  Inflammatory cytokines
Change in Functional Assessment of Cancer Therapy - Bone MarrowTransplantation (FACT-BMT) score | 8 weeks
  Assessment of Quality of Life
Change in General Sleep Disturbances Scale (GSDS) score | 8 weeks
  Assessment of sleep disturbance
Change in Global07, from PROMIS® Numeric Rating Scale v.1.0 - Pain Intensity 1a plus PAININ20, from PROMIS - Ca Item Bank v1.1 - Pain Interference score | 8 weeks
  Assessment of pain
Change in Hospital Anxiety and Depression Scale (HADS) score | 8 weeks
  Assessment of mood including anxiety and depression.
Change in the Godin Leisure Form (GLF) score | 8 weeks
  Assessment of physical activity

CONTACTS AND LOCATIONS:
Overall Officials: Nosha Farhadfar, MD, Principal Investigator — University of Florida; Wendy Dahl, PhD, Principal Investigator — University of Florida
Locations (1):
- Shands at University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided
Not yet determined.